CLINICAL TRIAL: NCT03389854
Title: Efficacy of Penile Traction Therapy Using a Novel Device: A Controlled, Single-blinded, Randomized Trial
Brief Title: Efficacy of Penile Traction Therapy Using a Novel Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Landon W. Trost, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-001283
Record Dates: First submitted 2017-10-19; First posted 2018-01-04 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Penile Diseases
MeSH Terms: conditions — Penile Diseases

STUDY DESIGN:
Intervention Model Description: Men will be randomized into one of four groups: no traction therapy, penile traction 30 minutes once daily, penile traction 30 minutes twice daily, and penile traction 30 minutes three times daily. This treatment will continue for 3 months, after which men will enter an open label phase for 3 months. Primary and secondary outcomes will be evaluated at the completion of the 3 month and 6 month time points. Additional AEs will be assessed at 9 months after study initiation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Objective outcomes including penile length and curvature will be masked for the investigator and outcome assessor by obtaining photographs of the penis in the lateral and dorsal planes. Curvatures will also be assessed by a clinician in the case where photographs are not able to be obtained or if the participant refuses photographs. These will be assessed without any knowledge as to which grouping the patient is located by two independent reviewers. If there are differences >5 degrees (curvature), or 0.5 cm (length), a 3rd individual will mediate the difference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Group 1 - Control (Sham Comparator): No treatment will be administered for the initial 3 months. This are is necessary as Peyronie's disease may result in changes in length and curvature as a function of the disease process. After the 3 month period of time, this group will enter an open label phase where they may utilize a penile traction device if desired.
  Interventions: Device: RestoreX PTT - open label phase only
- Group 2 - PTT 1x daily x 3 months (Experimental): Men will utilize penile traction therapy for 30 minutes once daily for the initial 3 months. After this phase is completed, they will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
  Interventions: Device: RestoreX PTT - randomized and open label
- Group 3 - PTT 2x daily x 3 months (Experimental): Men will utilize penile traction therapy for 30 minutes twice daily for the initial 3 months. After this phase is completed, they will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
  Interventions: Device: RestoreX PTT - randomized and open label
- Group 4 - PTT 3x daily x 3 months (Experimental): Men will utilize penile traction therapy for 30 minutes three times daily for the initial 3 months. After this phase is completed, they will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
  Interventions: Device: RestoreX PTT - randomized and open label

INTERVENTIONS:
Device: RestoreX PTT - randomized and open label — Penile traction therapy in the straight and bent positions
  Arms: Group 2 - PTT 1x daily x 3 months; Group 3 - PTT 2x daily x 3 months; Group 4 - PTT 3x daily x 3 months
Device: RestoreX PTT - open label phase only — Penile traction therapy in the straight and bent positions
  Arms: Group 1 - Control

SUMMARY:
This clinical trial is designed to assess the safety, dosing, and preliminary efficacy of a novel penile traction device on correcting deformities relating to Peyronie's disease, a condition which results in penile curvature and length loss. The trial is designed as a randomized, placebo-controlled study with men randomized to receiving no therapy or penile traction therapy 30 minutes once, twice, or three times daily. The study will occur over a 3 month period, after which an open label phase for 3 months will be conducted. Final assessments for adverse effects will also be assessed at 9 months.

DETAILED DESCRIPTION:
Peyronie's disease (PD) is a fibrotic condition of the penis, affecting 1-13% of the US male population. The disease results in penile curvature and significant psychosocial bother. Current preferred therapies for PD include repeated penile injections with bacterial enzymes and surgery. However, these therapies are expensive and in some cases result in permanent reductions in penile length and sensation. Penile traction therapy (PTT) is a relatively newer treatment which has been proposed as a treatment for PD with preliminary data suggesting a potential role. However, currently available PTT devices are primarily designed for penile lengthening and have many significant limitations including a requirement of use for 9 hours daily and significant difficulties in personal application. Given these limitations, a new penile traction device (RestoreX® ) was created and funded through Mayo Ventures and was specifically designed to treat men with PD. The primary objective of the current study is to evaluate safety of the device using various dosing schedules, with secondary endpoints designed to assess efficacy and subjective outcomes. To accomplish the study, a population of men from Mayo Clinic with PD will be enrolled and will be randomized to utilize the device for varying amounts of time. Outcomes will be assessed at 3, 6, and 9 months, and results are to be used with the intent to publish in a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Peyronie's disease
* Current 30 degree curvature in a single plane (i.e. 20 degrees up, 15 degrees left would not be a candidate)
* Not undergoing other therapies for PD currently

Exclusion Criteria:

* Stretched penile length <7 cm
* Prisoners
* Erectile dysfunction unresponsive to phosphodiesterase-5 inhibitors or intracavernosal injection therapies
* Diabetes mellitus with evidence of end-organ damage (peripheral neuropathy, retinopathy, chronic kidney disease stage III or higher)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Landon Trost, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joseph J, Ziegelmann MJ, Alom M, Savage J, Kohler TS, Trost L. Outcomes of RestoreX Penile Traction Therapy in Men With Peyronie's Disease: Results From Open Label and Follow-up Phases. J Sex Med. 2020 Dec;17(12):2462-2471. doi: 10.1016/j.jsxm.2020.10.003. Epub 2020 Nov 20. PMID 33223425
- [Derived] Ziegelmann M, Savage J, Toussi A, Alom M, Yang D, Kohler T, Trost L. Outcomes of a Novel Penile Traction Device in Men with Peyronie's Disease: A Randomized, Single-Blind, Controlled Trial. J Urol. 2019 Sep;202(3):599-610. doi: 10.1097/JU.0000000000000245. Epub 2019 Aug 8. PMID 30916626
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: No treatment will be administered for the initial 3 months. After the 3 month period of time, this group will enter an open label phase where they may utilize a penile traction device if desired.
- Penile Traction Therapy Group 1x Daily x 3 Months: Men will utilize penile traction therapy for 30 minutes once daily for the initial 3 months. After this phase is completed, they will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
- Penile Traction Therapy Group 2x Daily x 3 Months: Men will utilize penile traction therapy for 30 minutes twice daily for the initial 3 months. After this phase is completed, they will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
- Penile Traction Therapy Group 3x Daily x 3 Months: Men will utilize penile traction therapy for 30 minutes three times daily for the initial 3 months. After this phase is completed, they will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
Period: Overall Study
Arm/Group | Control Group | Penile Traction Therapy Group 1x Daily x 3 Months | Penile Traction Therapy Group 2x Daily x 3 Months | Penile Traction Therapy Group 3x Daily x 3 Months
Started | 28 | 27 | 28 | 27
Completed | 27 | 21 | 23 | 19
Not Completed | 1 | 6 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Penile Traction Therapy Group 1x Daily x 3 Months | Penile Traction Therapy Group 2x Daily x 3 Months | Penile Traction Therapy Group 3x Daily x 3 Months | Total
Number analyzed (Participants) | 28 | 27 | 28 | 27 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.7) | 56.6 (8.3) | 59.0 (6.9) | 60.0 (5.5) | 58.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 28 | 27 | 28 | 27 | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 28 | 27 | 110

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events at Baseline
Description: Percentage of participants being treated with penile traction to experience adverse events relating to device use defined by redness, pain, swelling, new bumps, discoloration, sensation loss, abnormal sensation or other
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Penile Traction Therapy Group 1x Daily x 3 Months | Penile Traction Therapy Group 2x Daily x 3 Months | Penile Traction Therapy Group 3x Daily x 3 Months
Number analyzed (Participants) | 27 | 28 | 27
percentage of participants
  Penile erythema or discoloration | 2 | 2 | 1
  Loss or abnormal penile sensation | 7 | 10 | 7

2. Primary Outcome: Adverse Events at 3 Months
Description: as for outcome 1
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Penile Traction Therapy Group 1x Daily x 3 Months | Penile Traction Therapy Group 2x Daily x 3 Months | Penile Traction Therapy Group 3x Daily x 3 Months
Number analyzed (Participants) | 27 | 28 | 27
percentage of participants
  Transient Erythema | 43 | 41 | 37
  Transient Sensory Changes | 10 | 14 | 16
  Transient Discomfort | 33 | 50 | 37

3. Primary Outcome: Adverse Events at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- Open Label Period Penile Traction Therapy: After the initial 3 month study period subjects from both the control group and the penile traction therapy group will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
Arm/Group | Open Label Period Penile Traction Therapy
Number analyzed (Participants) | 63
percentage of participants
  Penile erythema or discoloration | 35
  Loss or abnormal penile sensation | 5
  New penile pain, Mild | 27

4. Primary Outcome: Adverse Events at 9 Months
Description: as for outcome 1
Time Frame: 9 months
Measure: Number; unit: percentage of participants
Groups:
- Open Label Penile Traction Therapy: After the initial 3 month study period subjects from both the control group and the penile traction therapy group will enter an open label phase for 3 months where they may utilize the device as much or as little as desired.
Arm/Group | Open Label Penile Traction Therapy
Number analyzed (Participants) | 57
percentage of participants
  Penile erythema or discoloration | 4
  New penile pain, Mild | 4

5. Secondary Outcome: Change in Penile Length to Corona
Description: Stretched penile length measured in centimeters from pubic symphysis to glanular corona
Time Frame: 3 months, 6 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis. Data for 27 subjects control group and 62 subjects PTT group available for analysis at 3 mo. Data for 14 subjects original control group and 37 subjects original PTT group available for analysis at 6 mo.
Measure: Mean (Standard Deviation); unit: Centimeters
Groups:
- Penile Traction Therapy Group: RestoreX for 30 minutes (15 minutes straight and 15 minutes with counter bending) once, twice or 3 times daily as Penile Traction Therapy (PTT).
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 27 | 62
Centimeters
  3 month | 0.3 (0.8) | 1.3 (1.1)
  6 month: number analyzed (Participants) | 14 | 37
  6 month | 2.0 (1.1) | 2.3 (2.0)
Statistical Analysis 1: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs Penile Traction Therapy Group at 3 months; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs Penile Traction Therapy Group at 6 months; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Penile Length to Tip
Description: Stretched penile length measured in centimeters from pubic symphysis to penile tip
Time Frame: 3 months, 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 27 | 62
Centimeters
  3 months | 0.0 (0.7) | 1.5 (1.1)
  6 months: number analyzed (Participants) | 14 | 37
  6 months | 1.6 (1.2) | 1.9 (1.3)
Statistical Analysis 1: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs Penile Traction Therapy Group at 3 months; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs. Penile Traction Therapy Group at 6 months; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Penile Curvature
Description: Subjects received Trimix to achieve pharmacological erection and curvature was measured in degrees. A negative result denotes an improvement in curvature.
Time Frame: 3 months, 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 27 | 62
degrees
  3 months | 1.3 (19.0) | -11.7 (15)
  6 months: number analyzed (Participants) | 14 | 37
  6 months | -12.5 (18.6) | -14.9 (18.1)
Statistical Analysis 1: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs Penile Traction Therapy Group at 3 months; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs. Penile Traction Therapy Group at 6 months; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change Erectile Function
Description: Self reported International Index of Erectile Function (IIEF) questionnaire for erectile dysfunction (ED) scored on a scale of <11 severe ED, 11-16 moderate ED, 17-25 mild ED, 26-30 no ED. Questionnaires were given to participants at baseline, 3 months and 6 months. Change in the score was reported for 3 months and 6 months.
Time Frame: 3 months, 6 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis. Questionnaire 26 subjects control group and 59 subjects PTT group available for analysis 3 mo. Questionnaire 14 subjects original control group and 37 subjects original PTT group available for analysis 6 mo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 26 | 59
units on a scale
  3 months | -1.3 (6.7) | 2.5 (6.3)
  6 months: number analyzed (Participants) | 14 | 37
  6 months | 1.8 (4.4) | 4.4 (7.4)
Statistical Analysis 1: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs Penile Traction Therapy Group at 3 months; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control Group vs Penile Traction Therapy Group; Control group vs Penile Traction Therapy Group at 6 months; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Peyronie's Disease Psychological and Physical Domain on Peyronie's Disease Questionnaire (PDQ)
Description: Self reported Peyronie's Disease questionnaire (physical and psychological) severity score range 0 (none) to 4 (very severe) on 6 questions with a total score range 0 to 24. Negative denotes improvement.
Time Frame: Baseline, 3 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 23 | 59
units on a scale | -0.6 (3.3) | -2.3 (4.1)
Statistical Analysis 1: Comparison: Control Group vs Penile Traction Therapy Group; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Peyronie's Disease Penile Pain Domain on Peyronie's Disease Questionnaire (PDQ)
Description: Self reported Peyronie's Disease questionnaire penile pain scale range 0 (no pain) and 10 (extreme pain) on 3 questions with a total score range 0 to 30. Negative denotes improvement.
Time Frame: Baseline, 3 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 23 | 59
units on a scale | -0.8 (3.6) | -1.4 (3.2)
Statistical Analysis 1: Comparison: Control Group vs Penile Traction Therapy Group; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Peyronie's Disease Bother Domain of the Peyronie's Disease Questionnaire (PDQ)
Description: Self reported Peyronie's Disease questionnaire bother score range 0 (no issue or not at all bothered) and 4 (extremely bothered) on 4 questions with a total score range 0 to 16. Negative denotes improvement.
Time Frame: Baseline, 3 month
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 23 | 59
units on a scale | -0.9 (4.2) | -2.4 (3.4)
Statistical Analysis 1: Comparison: Control Group vs Penile Traction Therapy Group; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Overall Treatment Satisfaction
Description: Self reported satisfaction of penile traction therapy on a scale of very satisfied, somewhat satisfied, neutral, somewhat dissatisfied, very dissatisfied
Time Frame: 3 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Penile Traction Therapy Group
Number analyzed (Participants) | 63
percentage of participants
  % Very Satisfied | 25.4
  % Somewhat satisfied | 41.3
  % Neutral | 30.2
  % Somewhat dissatisfied | 3.2
  % Very dissatisfied | 0

13. Secondary Outcome: Ability to Achieve Sexual Intercourse
Description: Change from no to yes on the self reported standardized sexual encounter profile questions 2 "able to penetrate"
Time Frame: 3 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 24 | 48
percentage of participants | 0 | 4

14. Secondary Outcome: Satisfaction With the RestoreX® Device to Alternative Forms of PTT
Description: Self reported satisfaction with how RestoreX® compares to other devices on a scale of much better, somewhat better, equal, somewhat worse, much worse
Time Frame: 3 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Penile Traction Therapy Group
Number analyzed (Participants) | 15
percentage of participants
  % RestoreX is much better | 86.7
  % RestoreX is somewhat better | 13.3
  % Both are equal | 0
  % RestoreX is somewhat worse | 0
  % RestoreX is much worse | 0

15. Secondary Outcome: Satisfaction With the RestoreX® Device to Alternative PD Therapies
Description: Subjects being treated for PD the first time were asked which therapies they would choose. Respondents could select more than 1 option so values equal greater than 100%.
Time Frame: 3 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Penile Traction Therapy Group
Number analyzed (Participants) | 54
percentage of participants
  RestoreX | 74.1
  Collagenase clostridium histolyticum | 23.6
  Oral pills | 14.8
  Vacuum erection device | 5.6
  Surgery | 1.8
  Other therapy | 1.8
  Other traction device | 0

16. Secondary Outcome: Ability to Achieve Sexual Intercourse
Description: Change from no to yes on the self reported standardized sexual encounter profile questions 2 "able to penetrate"
Time Frame: 6 months
Population: It was pre-specified to combine Penile Traction Therapy Groups for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Penile Traction Therapy Group
Number analyzed (Participants) | 14 | 37
percentage of participants | 0 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 9 month period for each subject receiving penile traction therapy.
Arm/Group | Penile Traction Therapy Group 1x Daily x 3 Months | Penile Traction Therapy Group 2x Daily x 3 Months | Penile Traction Therapy Group 3x Daily x 3 Months | Open Label Period Penile Traction Therapy
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28 | 0/27 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/27 | 0/63
Other Adverse Events (participants affected / at risk) | 16/27 | 15/28 | 13/27 | 28/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Penile Traction Therapy Group 1x Daily x 3 Months (N=27) | Penile Traction Therapy Group 2x Daily x 3 Months (N=28) | Penile Traction Therapy Group 3x Daily x 3 Months (N=27) | Open Label Period Penile Traction Therapy (N=63)
Penile erythema or discoloration, transient (Reproductive system and breast disorders) | 12 (12) | 12 (12) | 10 (10) | 24 (24) — 3 month outcomes among men in PTT group
Loss or abnormal penile sensation, transient (new onset for 6-, 9-month cohorts) (Reproductive system and breast disorders) | 3 (3) | 4 (4) | 4 (4) | 3 (3) — Total includes men who either had symptom at 6 or 9 months
New penile pain, transient (mild) (Reproductive system and breast disorders) | 9 (9) | 14 (14) | 10 (10) | 19 (19) — At 3 month time point (among men treated with traction)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03389854/Prot_SAP_000.pdf